CLINICAL TRIAL: NCT05178394
Title: The Influence of Weightlifting Belts and Wrist Straps on Deadlift Kinematics, Time to Complete a Deadlift and Rating of Perceived Exertion in Male Recreational Weightlifters
Brief Title: Weightlifting Belts and Wrist Straps for Weightlifters
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Education University of Hong Kong (Other)
Responsible Party: Principal Investigator, Shirley S.M. Fong, Principal investigator, The University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 00001
Record Dates: First submitted 2021-11-20; First posted 2022-01-05 (Actual); Last update posted 2022-01-05 (Actual); Status verified 2021-12

CONDITIONS: Exercise Movement Techniques

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Male recreational weightlifters (Experimental)
  Interventions: Device: Weightlifting belts and wrist straps

INTERVENTIONS:
Device: Weightlifting belts and wrist straps — The participants wore a weightlifting belt (Heavywear Nylon Contour Belt H9, North Carolina, USA) for the "with weightlifting belt" conditions and/or put on a pair of wrist straps (Versa Gripps Professional Series, Versa Gripps, Maine, USA) for the "with wrist strap" conditions. The steps involved in completing a conventional deadlift have been detailed in Holmes.

SUMMARY:
Objective: This study examined the effects of weightlifting belts and wrist straps on the kinematics of the deadlift exercise, time to complete a deadlift and rating of perceived exertion (RPE) in male recreational weightlifters.

Methods: Twenty participants used various combinations of belt and straps during a conventional deadlift. The hip and knee flexion, cervical lordosis, thoracic kyphosis and lumbar lordosis angles and time to complete a deadlift were measured using video analysis software. RPE was also recorded.

ELIGIBILITY:
Inclusion Criteria:

* men
* aged 18 to 30 years
* more than 3 years of weightlifting experience
* have been training at least 4 hours per week
* engage in recreational weightlifting

Exclusion Criteria:

* musculoskeletal disorders (e.g., leg length discrepancies and severe flat feet)
* neurological disorders (e.g., epilepsy)
* spinal problems (e.g., scoliosis)
* upper limb problems (e.g., history of shoulder dislocation, tennis or golf elbow)
* recent injuries that could affect performance
* train regularly for other sports.

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 20 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
Hip flexion angle | Through study completion, an average of two hours
  Hip flexion angle during setup phase of a deadlift
Knee flexion angle | Through study completion, an average of two hours
  Knee flexion angle during setup phase of a deadlift
Cervical lordosis angle | Through study completion, an average of two hours
  Cervical lordosis angle during lockout phase of a deadlift
Thoracic kyphosis angle | Through study completion, an average of two hours
  Thoracic kyphosis angle during lockout phase of a deadlift
Lumbar lordosis angle | Through study completion, an average of two hours
  Lumbar lordosis angle during lockout phase of a deadlift

SECONDARY OUTCOMES:
Time | Through study completion, an average of two hours
  Time to complete a deadlift
Rating of perceived exertion | Through study completion, an average of two hours
  Rating of perceived exertion during a deadlift

CONTACTS AND LOCATIONS:
Locations (1):
- University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No
Confidentiality of participant information.